CLINICAL TRIAL: NCT00179829
Title: Detection of Minimal Residual Disease in Newly Diagnosed Patients With Leukemia and Those Who Undergo a Bone Marrow Transplant Using the Wilms Tumor Suppressor Gene (WT1) as a Marker By RT-PCR
Brief Title: WT1 for the Detection of Minimal Residual Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 0399
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Leukemia; Cancer
Keywords: leukemia; acute lymphocytic leukemia; chronic myelogenous leukemia; acute myelogenous leukemia
MeSH Terms: conditions — Leukemia; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute

INTERVENTIONS:
Procedure: WT 1 Testing

SUMMARY:
The purpose of this study is to determine if WT1 is an adequate measurement of minimal residual disease in leukemic patients.

DETAILED DESCRIPTION:
Patients with acute Leukemia may have a large number of leukemic cells at the time that leukemia is evident clinically. At the time that we determine that a patient is in complete remission (CR) the patient may still have leukemic cells present in smaller quantities. One of the most important factors in the successful treatment of patients with leukemia is the ability to determine if the eradication of leukemia has been achieved. The determination of Minimal Residual Disease may be important in the determination of the therapy that a given patient will receive as determined by the level of residual disease.

WT1 gene function and expression. The WT1 gene is a candidate gene for Wilms tumor, which is thought to arise as a result from inactivation of both alleles of the WT1 gene located at chromosome 11p13. The WT1 gene has been considered a tumor suppressor gene because intragenic deletions or mutations are found in tumors, germline mutations have been found in-patients with leukemia, and mediates growth suppression of Wilms tumor cells expressing a WT1 splicing variant.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 21 years of age.
* Patients with the following diseases: Acute lymphoblastic Leukemia (ALL) at the time of diagnoses or relapse, Acute non-lymphoblastic leukemia (ANLL) at diagnosis or after relapse and Chronic Myelogenous leukemia in chronic or accelerated phase.
* Patients will be eligible for any of the available treatment protocols or protocols for stem cell transplantation, regardless of the source of stem cells.
* Patients or legal guardians will sign an Institutional Review Board (IRB) approved informed consent.
* Patients will have venous access or peripheral vein for sampling.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 1999-02 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To assess the presence of the WT1 gene at the time of relapse in-patients with acute or chronic leukemia.
To determine longitudinally its value as a marker for minimal residual disease (MRD) and its correlation to leukemia free survival after bone marrow transplantation.
To assess the presence of the WT1 gene in newly diagnosed patients with leukemia (ALL, ANLL) at the time of diagnoses and during the course of their treatment and correlate it with leukemia free survival (LFS) and relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Morris Kletzel, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States